CLINICAL TRIAL: NCT05359692
Title: Phase 2, Open-Label, Multicenter Study of INCAGN01876 in Combination With Immunotherapy in Participants With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: INCAGN01876 in Combination With Immunotherapy in Participants With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision; no safety concerns
Sponsor: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCAGN 1876-204
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Advanced Malignancies; Recurrent Head and Neck Squamous Cell Carcinoma
Keywords: carcinoma; carcinoma, squamous cell; squamous cell carcinoma of head and neck; anti-PD-(L)1 therapy; HNSCC; SCCHN
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma; Carcinoma, Squamous Cell

STUDY DESIGN:
Masking Description: open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Cohort 1 (Experimental): INCAGN01876 every 2 weeks (Q2W) with retifanlimab every 4 weeks (Q4W).
  Interventions: Biological: INCAGN01876; Biological: retifanlimab
- Part 1: Cohort 2 (Experimental): INCAGN01876 Q2W with retifanlimab Q4W.
  Interventions: Biological: INCAGN01876; Biological: retifanlimab
- Part 2 (Expansion): Treatment Group A (Experimental): INCAGN01876 and retifanlimab combination in participants who have been previously treated with anti-PD-(L)1 therapy.
  Interventions: Biological: INCAGN01876; Biological: retifanlimab
- Part 2 (Expansion): Treatment Group B (Experimental): INCAGN01876 and retifanlimab combination in participants who are naive to anti-PD-(L)1 therapy.
  Interventions: Biological: INCAGN01876; Biological: retifanlimab

INTERVENTIONS:
Biological: INCAGN01876 — INCAGN1876 will be adminstered via IV at at the protocol-defined dose and schedule according to cohort and treatment group enrollment.
Biological: retifanlimab — retifanlimab will be administered via IV Q4W

SUMMARY:
The purpose of this study is to determine the safety, tolerability, efficacy, PK and pharmacodynamics of INCAGN01876 when given in combination with retifanlimab. The study will consist of 2 parts: a safety lead-in part (Part 1) followed by a dose expansion part (Part 2).

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety, tolerability, efficacy, PK and pharmacodynamics of INCAGN01876 when given in combination with retifanlimab in participants with GITR expression in recurrent or metastatic HNSCC who have progressed on or after prior systemic therapy including anti-PD-(L)1 therapy. The study will consist of 2 parts: a safety lead-in part (Part 1) followed by a dose expansion part (Part 2)

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent or metastatic HNSCC (oral cavity, oropharynx, hypopharynx, or larynx), that is not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy). Participants with squamous cell carcinomas of the nasopharynx, salivary gland, or nonsquamous cell histology are excluded.
* Documented progression on or after PD-(L)1 inhibitor alone or in combination with platinum-based chemotherapy for recurrent or metastatic HNSCC. Exception: Treatment Group B (Part 2, expansion): PD-(L)1-naïve.
* ECOG performance status of 0 to 1.
* Measurable disease based on RECIST v1.1.
* Mandatory pre-treatment and on-treatment tumor biopsies.
* GITR-positive tumor confirmed by central laboratory before study treatment start.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Have received chemotherapy, targeted small molecule therapy or curative radiation within 21 days of first dose of study drug; prior mAB for anticancer therapy other within 28 days of first dose of study drug; or investigational study drugs or devices within 28 days or five half-lives prior to enrollment unless approved by medical monitor.
* Prior treatment with any TNF Super Family agonist therapy.
* Have not recovered to ≤ Grade 1 from toxic effects of prior therapy.
* Laboratory and medical history parameters not within the Protocol-defined range before the first administration of study treatment.

Known active HBV or HCV, or Known to be seropositive for HIV.

* Have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Known active infections requiring systemic treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2025-01-11 (Estimated)

PRIMARY OUTCOMES:
Part 1: Participants With Treatment-Emergent Adverse Events (TEAEs) | Screening through 90 days after end of treatment, up to 24 months
  A TEAE is any adverse event (AE) either reported for the first time or worsening of a pre-existing event after the first dose of study treatment.
Objective response rate (ORR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Assessed every 8 weeks for 12 months, thereafter every 12 weeks up to the end of treatment, up to 24 months.
  Defined as the percentage of participants having complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Duration of response (DOR) based on RECIST v1.1 and mRECIST | Assessed every 8 weeks for 12 months, then every 12 weeks, up to 24 months.
  Defined as the time from the earliest date of disease response (CR or PR) until earliest date of disease progression or death due to any cause.
Disease control rate (DCR) based on RECIST v1.1 and mRECIST | Assessed every 8 weeks for 12 months, then every 12 weeks, up to 24 months.
  Defined as the percentage of participants having CR, PR, or stable disease (SD).
Progression-free survival (PFS) based on RECIST v1.1 and mRECIST | Assessed every 8 weeks for 12 months, then every 12 weeks, up to 24 months.
  Defined as the time from the start of combination therapy until the earliest date of disease progression or death due to any cause.
Part 2: Participants With Treatment-Emergent Adverse Events (TEAEs) | Screening through 90 days after end of treatment, up to 24 months
  A TEAE is any adverse event (AE) either reported for the first time or worsening of a pre-existing event after the first dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nawel Bourayou, MD, Study Director — Incyte Corporation
Locations (17):
- United States (17):
  - Uab Medicine-the Kirklin Clinic, Birmingham, Alabama
  - University of California San Diego Medical Center, Moores Cancer Center, La Jolla, California
  - Stanford University, Palo Alto, California
  - Toi Clinical Research, Whittier, California
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland-Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Prime, New York, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Providence Portland Med. Ctr, Portland, Oregon
  - Md Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - The Adult Outpatient Pavilion At Vcu, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency